CLINICAL TRIAL: NCT06483555
Title: Subjects With Advanced Basal-like Pancreatic Adenocarcinoma Treated With Gemcitabine, Erlotinib and Nab-paclitaxel (PANGEA) Versus Subjects With Classical Pancreatic Adenocarcinoma Treated With Triplet Standard of Care Therapy.
Brief Title: Basal-like PDAC Treated With Gemcitabine, Erlotinib, and Nab-paclitaxel
Acronym: PANGEA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2220
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Adenocarcinoma; Metastatic Pancreatic Cancer; Basal Cell Neoplasm
Keywords: safety; tolerability; efficacy; EGFR inhibitors; gemcitabine; nab-paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms, Basal Cell | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel; Erlotinib Hydrochloride; Leucovorin; Oxaliplatin; folfirinox; Fluorouracil; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PurIST Basal (Experimental): Subjects will be screened using the PurIST classifier and "basal-like" tumors will be assigned combination therapy with GnP and erlotinib.
  Interventions: Drug: Gemcitabine; Drug: Nab paclitaxel; Drug: Erlotinib
- PurIST Classical (Active Comparator): Subjects will be screened using the PurIST classifier and with classical tumors will be treated per standard of care on triplet therapy.
  Interventions: Drug: NALIRIFOX; Drug: Folfirinox

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2, intravenously on day 1 and day 15, for subjects with basal-like cell type pancreatic carcinoma.
  Other Names: Gemcitabine hydrochloride; FF 10832; LY188011; C9H11F2N3O4 - HCl
  Arms: PurIST Basal
Drug: Nab paclitaxel — 125 mg/m2 intravenously on day 1 and day 15 for subjects with basal-like cell type pancreatic carcinoma.
  Other Names: Abraxane
  Arms: PurIST Basal
Drug: Erlotinib — 50 mg per oral daily. for subjects with basal-like cell type pancreatic carcinoma.
  Other Names: Tarceva
  Arms: PurIST Basal
Drug: NALIRIFOX — Subjects with classical pancreatic adenocarcinoma will receive. NALIRIFOX is liposomal irinotecan with 5-fluorouracil/leucovorin and oxaliplatin. Dosing and plan will be decided by the treating physician.
  Other Names: A combination of liposomal irinotecan,5 fluorouracil /leucovorin and oxaliplatin.
  Arms: PurIST Classical
Drug: Folfirinox — Subjects with classical pancreatic adenocarcinoma will receive. Dosing and plan will be decided by the treating physician.
  Other Names: It is a combination of leucovorin calcium (folinic acid), fluorouracil, irinotecan hydrochloride, and oxaliplatin
  Arms: PurIST Classical

SUMMARY:
This study explores the best dose of the combination treatment for subjects with advanced unresectable or metastatic basal-like subtype pancreatic adenocarcinoma. For that reason, the safety, efficacy, and tolerability, as well as preliminary estimates of anti-tumor effects of low-dose epidermal growth factor receptor EGFR inhibitors in combination with bi-weekly gemcitabine/nab-paclitaxel (GnP) will be examined in subjects with advanced basal-like pancreatic adenocarcinoma.

The Purity Independent Subtyping of Tumors (PurIST) will determine the type of cancer either "basal type" or "classical". If cancer subtype-based first-line chemotherapy in combination with erlotinib will be safe and tolerable in subjects with advanced unresectable or metastatic pancreatic adenocarcinoma of the basal-like subtype as defined by PurIST, as well as provide a preliminary assessment of treatment response in basal-like subjects. This study will also follow a subset of subjects with classical subtypes that are treated per standard of care on oxaliplatin-based triplet chemotherapy.

DETAILED DESCRIPTION:
The standard of care chemotherapy for first-line advanced pancreatic adenocarcinoma is FOLFIRINOX, NALIRIFOX, or gemcitabine/nab-paclitaxel. However, multiple studies suggest that basal-like subtypes of pancreatic adenocarcinoma do not respond to FOLFIRINOX. Based upon existing retrospective analyses, the addition of epidermal growth factor receptor (EGFR) inhibitors such as erlotinib to gemcitabine and nab-paclitaxel suggest improved rates of response in subjects with basal-like pancreatic adenocarcinoma compared to FOLFIRINOX.

Subjects with a classical subtype will be treated on standard-of-care oxaliplatin-based triplet chemotherapy. Subjects with basal type will receive the erlotinib combination treatment. The purpose of this study is to find out the best dose of the erlotinib combination treatment. The erlotinib combination treatment is not FDA-approved. However, the combinations of erlotinib, gemcitabine, and nab-paclitaxel are both approved by the FDA for the treatment of pancreatic cancer. The standard of care treatments are both FDA-approved. All three drugs have been used in combination before in other clinical trials and a certain amount of safety data exists.

In the basal-like arm of this study, a two-stage utility of bayesian optimal interval ( U-BOIN) design will be used to evaluate the range of safe and admissible doses in Stage 1 and the optimal best dose (OBD) in Stage 2 basal subjects. After the determination of the OBD, an expansion cohort will be enrolled to obtain additional precision of the overall response rate (ORR). In total, 52 patients will be enrolled in the basal-like arm. Separately, 52 patients with "classical" tumors will be enrolled in a parallel arm and given standard-of-care oxaliplatin-based triplet chemotherapy (FOLFIRINOX or NALIRIFOX) to determine long-term outcomes including overall survival, objective response rate, and progression-free survival. This is to test the safety and effectiveness (how well a treatment works) of both treatments, depending on the cancer type.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent was obtained to participate in the study and HIPAA authorization for release of personal health information. Subjects is willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* The subject must consent to a mandatory pre-study biopsy if archival tissue is not available or sufficient.
* Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria:

* Disease is not measurable according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1
* Not having histological or cytological evidence/confirmation of metastatic pancreatic adenocarcinoma.
* Prior pancreatic-focused therapy.
* Brain metastasis diagnosed within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adverse Events per Common Terminology Criteria for Adverse Events (NCI-CTCAE) | First day of study treatment through the 28 days after last treatment
  Adverse Events (AEs) will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, in Phase I subjects with basal-like settings. The number of participants with adverse events (AE) will be reported.
  .
Dose-limiting toxicity (DLT) | Up to 28 days
  DLTs are defined using adverse events as at least possibly related to erlotinib administration in Phase I subjects. If an apparent DLT is clearly due to an underlying disease and is unrelated to the product infusion, then the investigator will specify that the event is not a DLT. Toxicities related to treatment and assessed Adverse Events per Common Terminology Criteria for Adverse Events (NCI-CTCAE) will be used for assessment.
  The safety evaluation period for dose-limiting toxicity (DLT) assessment and determination of optimal best dose (OBD) will encompass toxicities related to treatment with low-dose erlotinib when administered with bi-weekly gemcitabine/nab-paclitaxel starting on the day of treatment initiation through the end of treatment.
The objective response rate- basal-like pancreatic carcinoma | Up to 12 weeks
  The objective response rate in Stage 2 subjects with basal-like histology, treated with low-dose erlotinib at the OBD when administered with bi-weekly gemcitabine/nab-paclitaxel as defined as complete response (CR) + partial response (PR) as determined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST) 1.1 criteria. RECIST indicates if the subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall survival- classical metastatic pancreatic adenocarcinoma | 2 years
  Overall survival of subjects with classical metastatic pancreatic adenocarcinoma is defined as the length of time from the start of treatment until death.

SECONDARY OUTCOMES:
The number of Adverse Events (AEs) in subjects with basal like pancreatic carcinoma | First day of study treatment through the 28 days after last treatment
  The number of Adverse Events (AEs) in subjects with basal-like pancreatic carcinoma treated with low-dose erlotinib when administered with bi-weekly gemcitabine/nab-paclitaxel as defined by CTCAE v5.
Progression-free survival | 2 years
  Progression-free survival in subjects on low-dose erlotinib when administered with bi-weekly gemcitabine/nab-paclitaxel with basal-like metastatic pancreatic adenocarcinoma is defined as the length of time between the start of treatment until progression or death.
Overall survival in subjects with basal-like metastatic pancreatic adenocarcinoma | 2 years
  Overall survival in subjects with basal-like metastatic pancreatic adenocarcinoma on low-dose erlotinib when administered with bi-weekly gemcitabine/nab-paclitaxel is defined as the length of time from the start of treatment until death (basal-like arm only).
The objective response in subjects with classical pancreatic adenocarcinoma | Up to 12 weeks
  The objective response in subjects with classical pancreatic adenocarcinoma treated with standard-of-care triplet chemotherapy (FOLFIRINOX or NALIRIFOX) as defined as complete response (CR) + partial response (PR) as determined by RECIST 1.1 criteria.
The number of Adverse Events (AEs) in subjects with classical pancreatic adenocarcinoma | First day of study treatment through the 28 days after last treatment
  The number of Adverse Events (AEs) in subjects with classical pancreas carcinoma treated with standard-of-care triplet therapy as defined by CTCAE v5.0.
Progression-free survival (PFS) in subjects with classical pancreatic adenocarcinoma | 2 years
  Progression-free survival (PFS) after standard-of-care triplet chemotherapy (FOLFIRINOX or NALIRIFOX) in patients with classical metastatic pancreatic adenocarcinoma is defined as the length of time between the start of standard-of-care triplet therapy until progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Somasundaram, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials